CLINICAL TRIAL: NCT02520375
Title: Effects of Prebiotic Oral Healthcare Products as an Adjunct to Non-surgical Periodontal Therapy
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Allocation: Randomized | Masking: Double
Other Study IDs: s58074
Record Dates: First submitted 2015-07-01; First posted 2015-08-11 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Periodontitis
MeSH Terms: conditions — Periodontitis | interventions — Prebiotics

ARMS (2):
- Prebiotic (Experimental): This group will be administered a prebiotic mouthrinse and toothpaste
  Interventions: Other: Prebiotic
- Control (Placebo Comparator): This group will be administered a control mouthrinse and toothpaste
  Interventions: Other: Control

INTERVENTIONS:
Other: Prebiotic
  Arms: Prebiotic
Other: Control
  Arms: Control

SUMMARY:
The aim of this study is to determine the impact of a prebiotic toothpaste and mouthrinse in periodontitis patients as an adjunct to scaling and rootplaning.

DETAILED DESCRIPTION:
The aim of this study is to determine the impact of a prebiotic toothpaste and mouthrinse in periodontitis patients as an adjunct to scaling and rootplaning. Study design: this study will be a single centre (Department of Oral Health Sciences, University Hospitals Leuven), double blind, randomized, placebo controlled clinical trial. The randomization (by means of a computer program) and double blind design are thought to minimize the bias of the investigator and patients. Study population: adults, who consult at the department of Periodontology at the University Hospital Leuven and who fit the inclusion criteria will be asked to participate in this study.

ELIGIBILITY:
Inclusion Criteria:

* 40 patients
* ≥ 36 years of age

  - Page 4 of 4 [DRAFT] -
* No previous scaling and rootplaning
* Clinical diagnosis: severe generalized periodontitis characterized by the presence of > 14 affected teeth when > 14 teeth are present (if number of teeth present is < 14, 8-14 teeth need to be affected) with an attachment loss of > 6mm prior to initial non-surgical periodontal therapy.
* A minimum of 3 natural teeth in every quadrant
* Willing and able to give written informed consent

Exclusion Criteria:

* Patients with aggressive periodontitis or necrotizing periodontitis
* Patients who smoke
* Pregnant or lactating woman
* A history of diabetes, rheumatic fever, liver or kidney disease, neurological deficiencies, or use of medication which may affect periodontal tissue, (phenytoin, cyclosporin, nifedipine, chronic use of non-steroidal antiinflammatory drugs)
* Patients with poorly controlled diabetes
* Patients taking bisphosphonate mediation
* Patient who have taken systemic antibiotics 3 months prior to treatment

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Primary Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Pocket Probing Depth (PPD) at teeth with residual pockets | Baseline - 6 months
  Pocket probing depth measured with Merrit B prob